CLINICAL TRIAL: NCT02035605
Title: A Phase 1 Single-ascending and Multiple-ascending Dose, Safety, Tolerability and Pharmacokinetics Study of Subcutaneously Administered ALN-AT3SC in Healthy Adult Volunteers and Hemophilia A or B Patients (Moderate or Severe Hemophilia)
Brief Title: A Phase 1 Study of an Investigational Drug, ALN-AT3SC, in Healthy Volunteers and Hemophilia A or B Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ALN-AT3SC-001
Record Dates: First submitted 2014-01-13; First posted 2014-01-14 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2018-06

CONDITIONS: Hemophilia A; Hemophilia B
MeSH Terms: conditions — Hemophilia A; Hemophilia B

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ALN-AT3SC (Active Comparator)
  Interventions: Drug: ALN-AT3SC
- Sterile Normal Saline (0.9% NaCl) (Placebo Comparator)
  Interventions: Drug: Sterile Normal Saline (0.9% NaCl)

INTERVENTIONS:
Drug: ALN-AT3SC — Ascending doses of ALN-AT3SC by subcutaneous (sc) injection
  Arms: ALN-AT3SC
Drug: Sterile Normal Saline (0.9% NaCl) — Calculated volume to match active comparator
  Arms: Sterile Normal Saline (0.9% NaCl)

SUMMARY:
The purpose of this study is to determine the safety, tolerability, and pharmacokinetics of ALN-AT3SC in healthy volunteers and Hemophilia A or B patients.

ELIGIBILITY:
Inclusion Criteria:

Part A (SAD phase) inclusion:

* Healthy adult males aged 18 to 40 years inclusive at Screening.
* Subjects with adequate complete blood counts and liver function tests.
* Willing to provide written informed consent and willing to comply with study requirements.

Part B & C (MAD & MD phase) inclusion:

* Adult male hemophilia patients aged 18 to 65 years inclusive at Screening.
* Patients with adequate complete blood counts and liver function tests.
* Patients with moderate or severe, clinically stable hemophilia A or B (Factor VIII or Factor IX ≤5%).
* Willing to provide written informed consent and willing to comply with study requirements

Part D (MD Phase in patients with inhibitors) Inclusion:

* Same as Parts B/C
* A Bethesda inhibitor assay > 0.6 BU/mL

Exclusion Criteria:

Part A (SAD phase) exclusion:

* Subjects with a personal history and/or family history of venous thromboembolism (VTE)
* Subjects with a known co-existing thrombophilic disorder
* Subjects with a history of multiple drug allergies or history of allergic reaction to an oligonucleotide or GalNAc.
* Subjects with a history of serious mental illness that includes, but is not limited to schizophrenia, bipolar disorder, severe depression requiring hospitalization or pharmacological intervention.
* Subjects who have a clinically relevant history or presence of cardiovascular, respiratory, gastrointestinal, renal, hematological, lymphatic, neurological, musculoskeletal, genitourinary, immunological including osteoarthritis and other inflammatory diseases, dermatological including rash, eczema, dermatitis, or connective tissue diseases or disorders.

Part B & C (MAD & MD phase) exclusion:

* Patients with a current serious mental illness that, in the judgment of the Investigator, may compromise patient safety, ability to participate in all study assessments, or study integrity.
* Patients who have a clinically relevant history or presence of cardiovascular, respiratory, gastrointestinal, renal, neurological, inflammatory or other diseases that in the judgment of the investigator precludes their participation in the study.
* Patients with a known co-existing thrombophilic disorder
* Patients with a history of multiple drug allergies or history of allergic reaction to an oligonucleotide or GalNAc.
* Patients who are known to be HIV positive and have a CD4 count <400 cells/μL

Part D (MD Phase in patients with inhibitors) exclusion:

* Same as Parts B/C
* Patients who are known to be HIV positive and have a CD4 count <200 cells/μL

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2014-01-20 (Actual); Primary Completion 2017-07-20 (Actual); Study Completion 2017-07-20 (Actual)

PRIMARY OUTCOMES:
The safety of ALN-AT3SC evaluated by the proportion of subjects experiencing adverse events (AEs), serious adverse events (SAEs), dose-limiting toxicities (DLTs), and AEs leading to study drug discontinuation. | Part A (SAD phase): through day 56; Part B (MAD) phase: through Day 70; Part C (MD Phase) through Day 112; Part D (MD Phase in patients with inhibitors) through Day 112

SECONDARY OUTCOMES:
The pharmacokinetics (PK) of ALN-AT3SC as characterized by plasma PK profiles and urine samples. | Part A (SAD) phase: through day 56; Part B (MAD) phase: through Day 70; Part C (MD Phase) through Day 112; Part D (MD Phase in patients with inhibitors) through Day 112
The pharmacodynamic (PD) effect of ALN-AT3SC, evaluated by Plasma AT levels. | Part A (SAD) phase: through day 56; Part B (MAD) phase: through Day 70; Part C (MD Phase) through Day 112; Part D (MD Phase in patients with inhibitors) through Day 112
The pharmacodynamic (PD) effect of ALN-AT3SC, evaluated by Plasma TG. | Part A (SAD) phase: through day 56; Part B (MAD) phase: through Day 70; Part C (MD Phase) through Day 112; Part D (MD Phase in patients with inhibitors) through Day 112

CONTACTS AND LOCATIONS:
Overall Officials: Kate Madigan, MD, Study Director — Alnylam Pharmaceuticals
Locations (13):
- Clinical Trial Site, Pittsburgh, Pennsylvania, United States
- Bulgaria (3):
  - Clinical Trial Site, Plovdiv
  - Clinical Trial Site, Sofia
  - Clinical Trial Site, Varna
- Russia (3):
  - Clinical Trial Site, Kirov
  - Clinical Trial Site, Moscow
  - Clinical Trial Site, Saint Petersburg
- Switzerland (2):
  - Clinical Trial Site, Sankt Gallen
  - Clinical Trial Site, Zurich
- United Kingdom (4):
  - Clinical Trial Site, Glasgow
  - Clinical Trial Site, London
  - Clinical Trial Site, Manchester
  - Clinical Trial Site, Truro

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pipe SW, Lissitchkov T, Georgiev P, Mangles S, Hegemann I, Trinchero A, Chowdary P, Forbes A, Feng L, Menapace LA, Kichou S, Andersson S, Demissie M, Ragni MV. Long-term safety and efficacy of fitusiran prophylaxis, and perioperative management, in people with hemophilia A or B. Blood Adv. 2025 Mar 11;9(5):1147-1158. doi: 10.1182/bloodadvances.2024013900. PMID 39642315
- [Derived] Pasi KJ, Rangarajan S, Georgiev P, Mant T, Creagh MD, Lissitchkov T, Bevan D, Austin S, Hay CR, Hegemann I, Kazmi R, Chowdary P, Gercheva-Kyuchukova L, Mamonov V, Timofeeva M, Soh CH, Garg P, Vaishnaw A, Akinc A, Sorensen B, Ragni MV. Targeting of Antithrombin in Hemophilia A or B with RNAi Therapy. N Engl J Med. 2017 Aug 31;377(9):819-828. doi: 10.1056/NEJMoa1616569. Epub 2017 Jul 10. PMID 28691885